CLINICAL TRIAL: NCT04628416
Title: Evaluation of the PICO® Negative Pressure Dressing System on the Fibula Free Flap Donor Site's Skin Graft.
Acronym: PICOFLAP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RECHMPL20_0047; 2020-A00425-34 (Other: ANSM)
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Carcinomatous Resections; Violent Trauma
Keywords: fibula free flap; skin graft

STUDY DESIGN:
Intervention Model Description: Randomized controlled multicentered trial with blinded evaluation of the primary outcome, comparing 2 management techniques applied on the skin graft done on the donor sites of fibula free flaps.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (Experimental)
  Interventions: Device: PICO dressing
- Control (Other)
  Interventions: Device: Conventional dressing

INTERVENTIONS:
Device: PICO dressing — Use of a portative miniature negative pressure dressing system named PICO® on the split-thickness skin graft of fibula free flap donor sites
  Arms: Experimental arm
Device: Conventional dressing — use of a conventional dressing (parrafin gauze) on the split-thickness skin graft of fibula free flap donor sites
  Arms: Control

SUMMARY:
A fibula free flap can be used for the reconstruction of a mandible or a maxillar when the lack of bonne exceeds 3cm. This flap is made of the fibula bone, some muscle around, the fibular vascular pedicle and a skin paddle to reconstruct the gum. Once this flap has been taken and transposed on the face, the leg is closed with a split thickness skin graft to replace the skin paddle. But the healing on this site is often a problem: this is partly due to the high rate of early graft's loss due to local devascularization (3 to 55% of loss). The skin grafting is generally improved by the application of a dressing sewn and left in place during 5 to 7 days postoperative (standard method). This study will evaluate the efficiency of a portative miniature negative pressure dressing system named PICO® on the split-thickness skin graft of fibula free flap donor sites, compared to the standard method. A prospective randomized evaluation will be done, comparing the PICO® to a conventional dressing. The main aim of the study is the evaluation of the impact of this portative system on the healing of the skin grafted donor site, in terms of rate of skin take, time of healing, complications and medical costs. The patients will be seen preoperatively to decide on their inclusion in the protocol. They will be reviewed at day 10 to evaluate the engraftment and possible local complications on the donor site. They will then be reviewed at day 20 and day 30 and until complete healing. The follow up will be of 12 months maximum. A medical cost evaluation will be done comparing the costs generated by the care on the donor site in the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Any patient requiring a fibula free flap with skin paddle
* Theoretical need of a skin graft for the closure of the donor site (evaluated by the surgeon in charge of the patient at the time of inclusion) and performed at the same time as the fibula flap
* Signature of informed consent.

Exclusion Criteria:

* Contraindication to making a fibula free flap:

  * anesthetic contraindication,
  * atheroma in the leg arteries obstructing more than 60% of the arterial lumen (objectified by CT angiography of lower limbs)
* Contraindication to the setting up of a negative pressure therapy:

  * allergy to one of the PICO® components
  * infection in the donor area
  * cutaneous lesions of the lower limb preventing the placement of an occlusive dressing or making it impossible to seal the device
* No affiliation to a social security scheme.
* Minor or major patients who are protected or unable to give their consent (according to article L1121-8 of the Public Health Code (PHC))
* Pregnant or lactating women (according to article L1121-5 of the PHC)
* Vulnerable people (according to article L1121-6 of the PHC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of failure of skin grafting (surface on which the skin graft did not take) | on Day 10 postoperative (+/- 2 days)

SECONDARY OUTCOMES:
Delay between the day of the operation and the complete healing of the donor site of the fibula flap (in days) | Through complete healing, a maximum of 1 year
  ): complete epithelialization of the grafted site with disappearing crusts, this evaluation will be performed by the nurse at home with photos addressed to the doctor in charge of the patient. At the approach of complete healing the patient will be seen in consultation for the exact dating of the healing. If necessary, several close consultations will be conducted to evaluate the complete healing date within +/- 7 days
Rate of other surgery due to a problem on the skin grafted area. | Through complete healing, a maximum of 1 year
Tendon exposure rate evaluated at day 10 (+/- 2 days) and day 20 (+/- 2 days) by the surgeon during hospitalization or in consultation if the patient is discharged. | Day 10 (+/- 2 days) and day 20 (+/- 2 days)
Rate of infection of the grafted site at day 10 (+/- 2 days) and day 20 (+/- 2 days), evaluated by the surgeon during hospitalization or in consultation if the patient is discharged | Day 10 (+/- 2 days) and day 20 (+/- 2 days)
Evolution of the quality of life at 1 month postoperative (+/- 4 days) compared to preoperative (assessed by the Short Form-12 Health Survey Version 2 (SF-12v2)) | At 1 month after surgery
Rate of patients for whom during of hospitalization was lengthened exclusively due to a problem with the skin graft. (Duration of hospitalization) | At 12 months
Evaluation of patient discomfort related to the PICO® device or to the standard dressing (noise, bulk, dressing) during the first 7 postoperative days. This discomfort is measured by an EVA of 0 to 100 measuring the discomfort experienced. | day 10
Treatment tolerance evaluation, measured wtih rate of adverse reaction | Day 20
Cost-effectiveness ratio. The medical and non-medical costs will be collect on the case report form | At 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Marie DE BOUTRAY, Montpellier, France